CLINICAL TRIAL: NCT05524844
Title: The Role of the Microbiome and Notch Signaling in Esophageal Adenocarcinoma
Brief Title: The Microbiome, Bile Acids, and Notch in Barrett's Esophagus (BE)
Status: Completed | Type: Observational
Sponsor: Columbia University (Other)
Collaborators: Weill Medical College of Cornell University (Other); National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Julian A Abrams, MD, Associate Professor of Medicine and Epidemiology, Columbia University
Other Study IDs: AAAT2456; R01CA255298 (NIH)
Record Dates: First submitted 2022-08-30; First posted 2022-09-01 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Barrett Esophagus; Esophageal Adenocarcinoma
Keywords: Saliva; Microbiome
MeSH Terms: conditions — Barrett Esophagus; Adenocarcinoma Of Esophagus | interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Saliva Esophageal brushings Esophageal biopsies Gastric aspirate
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Control: Non-BE controls undergoing endoscopy for any indication who are on stable dose Proton Pump Inhibitors for the past month.
  Interventions: Other: Sample Collection; Other: Endoscopy results; Other: Dietary questionnaire
- Barrett's Esophagus: Patients scheduled for upper endoscopy for clinical purposes, with a history of histologically confirmed Barrett's esophagus (2 cm length); 40 with no history of dysplasia, and 40 with high grade dysplasia or esophageal adenocarcinoma.
  Interventions: Other: Sample Collection; Other: Endoscopy results; Other: Dietary questionnaire

INTERVENTIONS:
Other: Sample Collection — Saliva, gastric aspirate, and esophageal brushings and biopsies.
Other: Endoscopy results — Results from standard of care endoscopy (scheduled separate of study)
Other: Dietary questionnaire — Diet History Questionnaire (II)

SUMMARY:
The purpose of this study is to prospectively collect and analyze clinical data and biospecimens from a cohort of 100 patients without BE (20), with non-dysplastic BE (40), or with BE and high grade dysplasia (HGD) or EAC (40). The investigators will enroll 80 patients scheduled for upper endoscopy for clinical purposes, with a history of histologically confirmed BE (2 cm length); 40 with no history of dysplasia, and 40 with HGD or EAC. The investigators will also enroll 20 non-BE controls undergoing endoscopy for any indication who are on stable dose proton-pump inhibitors (PPI) for the past month. PPI therapy is standard of care for BE patients.

DETAILED DESCRIPTION:
The incidence of esophageal adenocarcinoma (EAC) has risen 10-fold over the past half century and continues to have a dismal prognosis. Known risk factors for EAC do not adequately explain these incidence trends; the rise in EAC cases began a decade before increases in the prevalence of both gastro-esophageal reflux disease and obesity. Over the past 50+ years, dramatic changes in the bacterial composition (or microbiome) of the upper gastrointestinal tract have also occurred. While prior work has shown correlations between the microbiome, BE, and EAC, there is a critical knowledge gap on mechanisms by which bacteria interact with the esophagus and potentially promote cancer. The investigators hypothesize that increased levels of the certain bile acids in gastroesophageal reflux fluid cause changes that lead to increased interaction between bacteria and the esophagus, which may promote the development of esophageal adenocarcinoma (EAC). The investigators will carry out a case-control study of patients with and without BE, dysplasia, or EAC. The investigators will focus on deoxycholic acid in gastro-esophageal refluxate and its association with Notch signaling in tissue and bacterial composition. The microbiome represents a novel and potentially modifiable risk factor for the development of BE and EAC. Elucidation of microbiome features and mechanisms that promote the development of EAC is a critical step that will lead to subsequent trials of antibiotics, probiotics, and other interventions targeted to altering the microbiome, with the goal of lowering the risk of this highly lethal malignancy.

ELIGIBILITY:
Inclusion Criteria:

All subjects:

* Scheduled for an upper endoscopy
* Taking stable dose of a proton pump inhibitor at least once daily for 1 months prior to enrollment
* Eighteen years of age or older
* Able to give informed consent

Barrett's esophagus subjects only:

* Histologically confirmed BE (defined as endoscopically- suspected BE with intestinal metaplasia with goblet cells on esophageal biopsies)
* Maximal BE length ≥ 2 cm (Prague criteria: any C, M≥2)

Exclusion Criteria:

All subjects:

* History of head and neck cancer or esophageal or gastric cancer (except esophageal intramucosal adenocarcinoma)
* History of esophageal or gastric surgery
* Use of antibiotics or immunosuppressants within 1 month prior to endoscopy

Barrett's esophagus subjects only:

• History of prior endoscopic therapy for BE, except a history of prior endoscopic mucosal resection (EMR) of focal lesions withoutsubsequent ablative therapy is permitted

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study population will be based on the population of BE and EAC as well as the demographics of those who undergo upper endoscopy for other indications (the control population) at Columbia and Cornell, together with data drawn from numerous prior studies in our BE population.
Sampling Method: Non-Probability Sample
Enrollment: 54 (Actual)
Dates: Start 2021-02-09 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Concentration of Deoxycholic Acid (DCA) | 2 years
  To determine whether refluxate deoxycholic acid (DCA) is associated with increased Notch signaling in the development of esophageal adenocarcinoma (EAC), the investigators will calculate Pearson's correlation coefficients to assess within individual correlations between DCA and NOTCH3 gene expression.
Correlation between Enterobacteriaceae (from 16S) and NOTCH3 expression in BE tissue. | 2 years
  The within-individual correlation will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Julian Abrams, MD, Principal Investigator — Columbia University
Locations (2):
- United States (2):
  - Columbia University Irving Medical Center, New York, New York
  - Weill Cornell Medical Center, New York, New York

IPD SHARING:
Plan to Share IPD: No